CLINICAL TRIAL: NCT00204360
Title: Pediatric Epilepsy Database
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Other Study IDs: pediatric epilepsy database
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2005-08

CONDITIONS: Epilepsy
Keywords: epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
The purpose of this database is to collect information for clinical purposes on all children being treated for seizure disorders.

DETAILED DESCRIPTION:
At some point this information may be used to retrospectively review trends in seizure types, diagnostic evaluation and treatment (medical or surgical). The potential data recorded will be that of standard of care provided to these patients, including age, gender, seizure type/classification, diagnostic procedures (eg. EEG, MRI Magnetoencephalography {MEG}, Single Photon Emission Computed Tomography {SPECT}, Positron Emission Tomography {PET}, invasive electrocorticography) and various treatments (medications, diet, or neurosurgical interventions for the treatment of epilepsy). Records in the database will have identifiable information (name, date of birth, date of procedure, medical record number), but these identifying data will be removed, and only nonidentifying data will be used in the event of research completed using information from this clinical database.

ELIGIBILITY:
Inclusion Criteria:

* NONE

Exclusion Criteria:

* NONE

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Pongkiat Kankirawatana, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Children's Hospital of Alabama, Birmingham, Alabama, United States